CLINICAL TRIAL: NCT03891238
Title: Avelumab as Single Agent in Metastatic or Locally Advanced Urothelial Cancer in Patients Unfit for Cisplatin
Brief Title: Avelumab as Single Agent in Metastatic or Locally Advanced Urothelial Cancer in Patients Unfit for Cisplatin. The ARIES Study
Acronym: ARIES
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Consorzio Oncotech (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARIES
Record Dates: First submitted 2019-03-25; First posted 2019-03-26 (Actual); Last update posted 2024-02-01 (Actual); Status verified 2024-01

CONDITIONS: Metastatic or Locally Advanced PD-L1 Positive Urothelial Cancer
Keywords: unfit for cisplatin; PD-L1; urotelian metastatic cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — avelumab

STUDY DESIGN:
Intervention Model Description: To assess the activity of avelumab in patients with metastatic or locally advanced PD-L1 positive urothelial cancer not eligible for cisplatin-based chemotherapy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avelumab Arm (Experimental): Patients will receive avelumab at standard dosage of 10 mg/kg as a 1-hour intravenous infusion once every 2 weeks (Q2W).
  Interventions: Drug: Avelumab

INTERVENTIONS:
Drug: Avelumab — Patients will receive avelumab at standard dosage of 10 mg/kg as a 1-hour intravenous infusion once every 2 weeks (Q2W).

SUMMARY:
This is a single arm, open label, phase II study to evaluate the activity of avelumab (MSB0010718C) in patients with metastatic or locally advanced urothelial cancer considered unfit to cisplatin-based chemotherapy, to be conducted in conformance with Good Clinical Practices.

Cisplatin-unfit patients will be defined if at least one of these characteristics is present:

1. ECOG-Performance status = 2;
2. Creatinine Clearance < 60 ml/min;
3. Grade 2 or worse peripheral neuropathy or hearing loss;
4. Previous treatment with cisplatin for adjuvant intent in six months before the progression of disease.

DETAILED DESCRIPTION:
Each subject will participate in the trial from the time the subject signs the Informed Consent Form (ICF) through the final contact. After a screening phase of 28 days, each subject will receive the treatment. Treatment on trial will continue until disease progression is confirmed by the investigator/site radiologist, unacceptable adverse event(s), intercurrent illness that prevents further administration of treatment, investigator's decision to withdraw the subject, subject withdrawals consent, pregnancy of the subject, noncompliance with trial treatment or procedures requirements, or administrative reasons.

The study treatment may be continued after radiological progression of disease at physician discretion and if improvement of symptoms or not new symptoms were reported by the patient despite the radiological progression of disease.

Subjects who attain a complete response may consider stopping trial treatment if they meet criteria for holding therapy.

After the end of treatment given the potential risk for delayed immune-related toxicities, safety follow-up must be performed up to 90 days after the last dose of avelumab administration.

The extended safety follow-up beyond 30 days after last study drug administration may be performed either via a site visit or via a telephone call with subsequent site visit requested in case any concerns noted during the telephone call.

Subjects who discontinue for reasons other than disease progression will have post-treatment follow-up every 12 weeks for disease status until disease progression is confirmed by the investigator/site radiologist, initiating a non-study cancer treatment, withdrawing consent, or becoming lost to follow-up. All subjects will be followed by telephone for overall survival every 12 weeks until death, withdrawal of consent, or the end of the trial.

ELIGIBILITY:
Inclusion Criteria:

* • Be able to understand and be willing to sign a written informed consent for the trial. Informed consent obtained before any study-specific procedures.

  * Be Male or female patient ≥18 years of age on day of signing informed consent.
  * Have histologicallly or cytologically-confirmed diagnosis of urothelial cancer of the renal pelvis, ureter, bladder, or urethra. Both transitional cell and mixed transitional/non-transitional cell histologies are allowed, but transitional cell carcinoma must be the predominant histology. Subjects with non-urothelial cancer of the urinary tract are not allowed.
  * Have measurable or non-measurable disease according to Response Evaluation Criteria in Solid Tumors criteria (RECIST), version 1.1.
  * Have immunohistochemical expression of PD-L1 ≥ 5% on tumor cells in archived tumor biopsies.
  * Have a performance status of ≤2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale, as assessed within 10 days prior to treatment initiation.
  * Have a life expectancy of at least 6 months.
  * Female subject of childbearing potential and men must agree to use adequate contraception since signing of the informed consent form until at least 3 months after the last study drug administration. The investigator or a designated associate is requested to advise the subject how to achieve an adequate birth control. Highly effective contraception for both male and female subjects throughout the study and for at least 30 days after last avelumab treatment administration if the risk of conception exists. Adequate contraception is defined in the study as any medically recommend method (or combination of methods) as per standard of care.
  * Respect the Cisplatin-unfit criteria, defined if at least one of these characteristics is present:
* 1. ECOG-Performance status = 2;
* Creatinine Clearance < 60 ml/min;
* Grade 2 or worse peripheral neuropathy or hearing loss;
* Previous treatment with cisplatin for adjuvant intent in six months before the progression of disease.

  • Demonstrate adequate bone-marrow, liver, and renal function as assessed by the following laboratory requirements conducted within 7 days of starting to study treatment:
* Absolute neutrophil count (ANC) ≥ 1.5 × 109/L, platelet count ≥ 100 × 109/L, and hemoglobin ≥ 9 g/dL (may have been transfused);
* Total bilirubin ≤1∙5 × the upper limit of normal (ULN); or Direct bilirubin < ULN for subjects with total bilirubin levels >1.5xULN;
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST), levels ≤ 2.5 × ULN or AST and ALT levels ≤ 5 x ULN (for subjects with documented metastatic disease to the liver);
* International normalized ratio (INR) and partial thromboplastin time (PTT) ≤1∙5 × ULN. Subjects who are therapeutically treated with an agent such as warfarin or heparin will be allowed to participate if no prior evidence of an underlying abnormality in coagulation parameters exists. Close monitoring of at least weekly evaluations will be performed until INR and PTT are stable based on a pre-dose measurement as defined by the local standard of care;
* Platelet count ≥100.000/mm3, hemoglobin >9 g/dl, absolute neutrophil count >1.500/mm3;
* Alkaline phosphatase limit ≤2∙5 × ULN (≤5 × ULN for patients with liver metastases).
* Estimated creatinine clearance ≥ 30 mL/min according to the Cockcroft-Gault formula (or local institutional standard method);
* Pregnancy test: negative serum or urine pregnancy test at screening for women of childbearing potential.

Exclusion Criteria:

* • Has disease that is suitable for local therapy administered with curative intent.

  * Has received prior treatment with avelumab.
  * Has received prior therapy with an anti-PD-1 or anti-PD-L1 agent, or with an agent directed to another co-inhibitory T-cell receptor (e.g. CTLA-4, OX-40, CD137).
  * Known prior severe hypersensitivity to investigational product or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v 5.0 Grade ≥ 3).
  * Has received previous treatment for metastatic or locally advanced urothelial cancer.
  * Has a known previous or concurrent malignancy that is progressing or requires active treatment and is distinct in primary site or histology from urothelial cancer within 5 years before randomization.

Exceptions cervical cancer in situ or basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy. A history of prostate cancer that was identified incidentally following cystoprostatectomy for bladder cancer is acceptable, provided that the following criteria are met:

* Stage T2N0M0 or lower;
* Gleason score ≤ 6,
* PSA undetectable.

  * Has major surgical procedure, open biopsy, or significant traumatic injury within 28 days before start of study medication
  * Has active cardiac disease, defined as:

    1. Myocardial infarction or unstable angina pectoris within 6 months of the first date of study therapy.
    2. History of serious ventricular arrhythmia (i.e., ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring anti-arrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
    3. New York Heart Association (NYHA) Class III or greater congestive heart failure, or left ventricular ejection fraction of < 40%.
  * Has uncontrolled hypertension (systolic blood pressure >150 mmHg or diastolic pressure >90 mmHg despite optimal medical management)
  * Has arterial or venous thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), pulmonary embolism within the 4 months before start of study medication.
  * Persisting toxicity related to prior therapy (NCI CTCAE v. 5.0 Grade > 1); however, alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable
  * Active infection higher than National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0 grade 2 requiring systemic therapy.
  * Known history of testing positive for HIV or known acquired immunodeficiency syndrome.
  * Hepatitis B virus (HBV) or hepatitis C virus (HCV) infection at screening (positive HBV surface antigen or HCV RNA if anti-HCV antibody screening test positive).
  * Has seizure disorder requiring medication.
  * Vaccination within 4 weeks of the first dose of avelumab and while on trials is prohibited except for administration of inactivated vaccines
  * Has known symptomatic metastatic central nervous system (CNS) and/or meningeal tumors. Subjects with previously treated brain metastases may partecipate provided they are stable (the patient is >2 months from definitive therapy, has a negative imaging study within 4 weeks of study entry and is clinically stable - any neurologic symptoms have returned to baseline - with respect to the tumor at the time of study entry). Also, the patient must not be undergoing acute steroid therapy or tapering (chronic steroid therapy is acceptable provided that the dose is stable for 1 month before and after screening radiographic studies). This exception does not include carcinomatous meningitis, which is excluded regardless of clinical stability.
  * Has a history of organ allograft.
  * Has evidence or history of bleeding diathesis. Any hemorrhage or bleeding event of CTCAE grade 3 or higher within 4 weeks of start of study medication.
  * Has non-healing wound, ulcer, or bone fracture.
  * Has renal failure requiring hemodialysis or peritoneal dialysis.
  * Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. The use of physiologic doses of corticosteroids may be approved after consultation with the Sponsor.
  * Active autoimmune disease that might deteriorate when receiving an immuno-stimulatory agent. Patients with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
  * Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
  * Dehydration of NCI-CTCAE version 5.0 grade 1 or higher.Prior organ transplantation including allogenic stem-cell transplantation.
  * Non-healing wound, ulcer, or bone fracture.
  * Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
  * Has a history of substance abuse or medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
  * Has illness or medical conditions that are unstable or could jeopardize the safety of the patient and his or her compliance in the study.
  * Has interstitial lung disease with ongoing signs and symptoms at the time of informed consent.
  * Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2019-02-06 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Efficacy Endpoints | 2years
  This study aims to evaluate the anti-tumor efficacy of avelumab in patients with metastatic or locally advanced PD-L1 positive urothelial cancer not eligible for cisplatin-based chemotherapy.
  Overall Survival (OS) is the best endpoint to demonstrate the efficacy of antineoplastic immunotherapy.
  OS is defined as the time from study entry to the date of death (whatever the cause). The survival time of living patients will be censored at last date on which the patient is known to be alive or lost to follow-up. Subject status will be followed every 2 weeks while on treatment and then every 3 months thereafter.

SECONDARY OUTCOMES:
Median Progression-Free Survival (mPFS) | 18 months
  • mPFS: calculated from the date of study entry (first administration of avelumab) to date of documented radiographic progression or death according to RECIST Version 1.1 criteria.
  The primary analyses of PFS will be based on investigator's assessments using RECIST 1.1 criteria.
Objective response rate (ORR) | 18 months
  • ORR: defined as complete response (CR) or partial response (PR) according to RECIST Version 1.1 criteria as determined by investigator's assessments, obtained from start of study drug until documented radiographic disease progression.
  The first on study radiographic imaging assessment will be performed at 8 weeks (± 7 days) after first dose of study treatment and then every 12 weeks (± 7 days) thereafter or more frequently if clinically indicated.
  PR are those with greater than or equal to 30 percent decrease in the sum of the products of diameters (SOPD) of index lesions compared to the baseline SOPD, with no evidence of progressive disease (PD).
Safety Endpoints | 2 years
  The primary safety analysis will be based on subjects who experienced toxicities as defined by National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE), version 5.0 criteria. Safety will be assessed by quantifying the toxicities and grades experienced by subjects who have received avelumab, including serious adverse events (SAEs) and events of clinical interest (ECIs). Safety will be assessed by reported adverse events (AEs) according to NCI CTCAE version 5.0.
Patient Reported Outcomes (PRO) | 2 years
  The study aims to evaluate the quality of life assessed by EuroQoL EQ-5D. The eEuroQol-5D (eEQ-5D) is a standardized instrument for use as a measure of health outcome. The eEQ-5D will provide data for use in economic models and analyses including developing health utilities or QALYs. The five health state dimensions in this instrument include the following: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension is rated on a three-point scale from 1 (extreme problem) to 3 (no problem). The eEQ-5D also includes a graded (0 to 100) vertical visual analog scale on which the patient rates his or her general state of health at the time of the assessment. The eEQ-5D is to be completed at various time points as specified in the study Flow Chart, beginning with Cycle 1 until 30 days post-treatment discontinuation.

OTHER OUTCOMES:
Exploratory Objective(s) | 2 years
  Exploratory analysis will evaluate the predictive/prognostic role of the immunohistochemical expression of PD1/PD-L1 in tumor tissue samples of subjects with recurrent/progressive metastatic urothelial cancer not eligible for cisplatin-based chemotherapy and treated with avelumab.

CONTACTS AND LOCATIONS:
Locations (21):
- Italy (21):
  - Istituto Tumori "Giovanni Paolo II" IRCCS Ospedale Oncologico di Bari, Bari
  - ASST Papa Giovanni XXIII, Bergamo
  - Ospedale Santa Croce - A.O. Ospedali Riuniti Marche Nord, Fano
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Ospedale di Macerata - ASUR - Area Vasta N°3, Macerata
  - Istituto Europeo di Oncologia, Milan
  - Grande Ospedale Metropolitano Niguarda, Milan
  - INT- IRCCS - Foundation G. Pascale, Napoli
  - AOU San Luigi Gonzaga, Orbassano
  - Azienda Ospedaliera Universitaria di Parma, Parma
  - Fondazione Salvatore Maugeri, Pavia
  - A.O. Ospedali Riuniti Marche Nord, Pesaro
  - Azienda Ospedalieo-Universitaria Pisana, Pisa
  - Arcispedale Santa Maria Nuova Di Reggio Emilia, Reggio Emilia
  - Policlinico Universitario Campus Bio Medico, Roma
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma
  - Ospedale "S. Vincenzo" di Taormina, Taormina
  - Azienda Ospedaliera Santa Maria, Terni
  - Presidio Ospedaliero "Santa Maria Della Misericordia" Di Udine Sede Di Udine, Udine
  - Az.Osp.Universitaria Integrata Verona- Borgo Trento, Verona
  - ULSS 8 Berica- Ospedale San Bortolo di Vicenza, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Agata Y, Kawasaki A, Nishimura H, Ishida Y, Tsubata T, Yagita H, Honjo T. Expression of the PD-1 antigen on the surface of stimulated mouse T and B lymphocytes. Int Immunol. 1996 May;8(5):765-72. doi: 10.1093/intimm/8.5.765. PMID 8671665
- [Background] Ishida Y, Agata Y, Shibahara K, Honjo T. Induced expression of PD-1, a novel member of the immunoglobulin gene superfamily, upon programmed cell death. EMBO J. 1992 Nov;11(11):3887-95. doi: 10.1002/j.1460-2075.1992.tb05481.x. PMID 1396582
- [Background] Blank C, Brown I, Peterson AC, Spiotto M, Iwai Y, Honjo T, Gajewski TF. PD-L1/B7H-1 inhibits the effector phase of tumor rejection by T cell receptor (TCR) transgenic CD8+ T cells. Cancer Res. 2004 Feb 1;64(3):1140-5. doi: 10.1158/0008-5472.can-03-3259. PMID 14871849
- [Background] Dong H, Strome SE, Salomao DR, Tamura H, Hirano F, Flies DB, Roche PC, Lu J, Zhu G, Tamada K, Lennon VA, Celis E, Chen L. Tumor-associated B7-H1 promotes T-cell apoptosis: a potential mechanism of immune evasion. Nat Med. 2002 Aug;8(8):793-800. doi: 10.1038/nm730. Epub 2002 Jun 24. PMID 12091876
- See also: ARIES trial — https://www.oncotech.org/aries/